CLINICAL TRIAL: NCT06913062
Title: Combining Neural Mobilization With Conventional Rehabilitation: A New Approach to Cervico-Brachial Neuralgia Management
Brief Title: Neural Mobilization in Cervico-Brachial Neuralgia
Acronym: NM-CBN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, Selma Bouden, assistant doctor, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECR-OMG-2024-302; ECR-OMG-2024-303 (Other: Charles Nicolle Hospital)
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cervico Brachialgia
Keywords: cervico-brachial neuralgia; neural mobilization; pain; function
MeSH Terms: conditions — Brachial Plexus Neuritis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): For control group, the conventional rehabilitation protocol aimed to alleviate muscular and neuropathic pain in the short term, improve cervical mobility, reduce muscle tension, and increase muscle strength in the medium term, and promote a healthy lifestyle along with socio-professional reintegration in the long term. The principles included educating patients about their condition, respecting pain thresholds, and considering fatigue levels. Each patient received treatment for two months, with three sessions per week, each lasting about one hour. The protocol consisted of three phases: the first week focused on relaxation through massage and low-frequency electrotherapy; the second week introduced passive joint mobilizations; and from the third week, muscle stretching and strengthening exercises were incorporated. Additionally, functional exercises targeting daily activities and body awareness techniques are included to maintain proper posture.
  Interventions: Procedure: conventional rehabilitation
- NM arm (Experimental): For NM group, long-term goals included improving neuromeningeal mobility and restoring function to neural structures. Each patient received the treatment for two months, with three sessions per week, each lasting about one hour. After addressing joint limitations and muscle tensions affecting radicular mobility, NM was introduced starting from the fourth week. The protocol was structured around three main axes: treatment of interfaces (joint mobilizations and traction), direct treatment (using neurodynamic techniques), and indirect treatment (neural self-mobilization and lifestyle advice). The treatment included various stages for each ULNT technique [9]. ULNT1 targeted the median nerve and involved shoulder abduction, elbow extension, and head inclination. ULNT2 focused on scapular depression and targeted cervical roots. ULNT3 emphasized radial nerve tension with internal rotation of the shoulder, while ULNT4 addressed ulnar nerve tension through elbow flexion and shoulder abduction
  Interventions: Procedure: conventional rehabilitation; Procedure: neural mobilisation

INTERVENTIONS:
Procedure: conventional rehabilitation — For control group, the conventional rehabilitation protocol aimed to alleviate muscular and neuropathic pain in the short term, improve cervical mobility, reduce muscle tension, and increase muscle strength in the medium term, and promote a healthy lifestyle along with socio-professional reintegration in the long term. The principles included educating patients about their condition, respecting pain thresholds, and considering fatigue levels. Each patient received treatment for two months, with three sessions per week, each lasting about one hour. The protocol consisted of three phases: the first week focused on relaxation through massage and low-frequency electrotherapy; the second week introduced passive joint mobilizations; and from the third week, muscle stretching and strengthening exercises were incorporated. Additionally, functional exercises targeting daily activities and body awareness techniques are included to maintain proper posture.
Procedure: neural mobilisation — The protocol was structured around three main axes: treatment of interfaces (joint mobilizations and traction), direct treatment (using neurodynamic techniques), and indirect treatment (neural self-mobilization and lifestyle advice). The treatment included various stages for each ULNT technique. ULNT1 targeted the median nerve and involved shoulder abduction, elbow extension, and head inclination. ULNT2 focused on scapular depression and targeted cervical roots. ULNT3 emphasized radial nerve tension with internal rotation of the shoulder, while ULNT4 addressed ulnar nerve tension through elbow flexion and shoulder abduction. Each technique was executed with specific movements, maintained for 20 to 30 seconds, and repeated 15 times, followed by gentle scapular mobilizations until pain resolution.
  Arms: NM arm

SUMMARY:
This study aimed to compare the effectiveness of neural mobilization (NM) combined with conventional rehabilitation versus conventional rehabilitation alone in patients with chronic common cervico-brachial neuralgia (CBN), focusing on pain, cervical range of motion (ROM), functional disability, and psychological state.

A randomized controlled trial was conducted including patients with chronic CBN. They were randomized into two groups: control group received standard rehabilitation, while NM Group received the same treatment with additional NM techniques. Evaluations were conducted pre- and post-treatment, assessing pain, cervical ROM, functional disability and psychological state via the Beck Depression Inventory.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* with chronic common CBN

Exclusion Criteria:

* secondary CBN
* prior cervical surgery
* cervical trauma
* recent central or peripheral neurological conditions
* unstable cauda equina lesions,
* untreated tumors or infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | Outcome measures were collected at baseline prior to the intervention (T0) and at the end of the treatment period (T1).
  Pain: was assessed using the Visual Analog Scale (VAS) which ranges from 0 (no pain) to 10 (maximal imaginable pain)

SECONDARY OUTCOMES:
mobility | Outcome measures were collected at baseline prior to the intervention (T0) and at the end of the treatment period (T1).
  Joint mobility assessment: focused on both the qualitative and quantitative aspects of movement. Following active movement, the therapist conducts a passive evaluation to analyze the end-range of motion (ROM) and any associated pain
function | Outcome measures were collected at baseline prior to the intervention (T0) and at the end of the treatment period (T1).
  Functional assessment: was performed using the Copenhagen Neck Functional Disability Scale (CNFDS) in its Arabic version. It is a self-administered questionnaire that measures functional disability levels in patients suffering from cervical pain. The CNFDS consists of 15 questions addressing various aspects of daily life, including headache, sleep quality, concentration, and psychosocial factors such as social interaction and emotional relationships. Scores on the scale range from 0 (no disability) to 30 (maximum disability)
depression | Outcome measures were collected at baseline prior to the intervention (T0) and at the end of the treatment period (T1).
  Psychological evaluation: was conducted using the Beck Depression Inventory (BDI). The Arabic validated version of this inventory was used to gauge the psychological state of patients, providing a quantitative estimate of depressive symptoms. The BDI includes 21 items that describe specific behavioral manifestations of depression, rated on a scale from 0 to 3. The final score is interpreted in terms of depression severity: 0-9 indicates minor depression, 10-18 indicates mild depression, 19-29 indicates moderate depression, and 30-63 indicates severe depression

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Nicolle Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No